CLINICAL TRIAL: NCT06399666
Title: Impact of Inflammatory Indexes and Gene Scores in Prediction of Atrial Fibrillation - IERV Trial
Brief Title: Impact of Inflammatory Indexes and Gene Scores in Prediction of Atrial Fibrillation
Acronym: IERV
Status: Recruiting | Type: Observational
Sponsor: Vrinnevi Hospital (Other)
Collaborators: Ryhov County Hospital (Other)
Responsible Party: Principal Investigator, Jakob Hytting, MD, Department of Cardiology, Principal Investigator, Doctoral Candidate, Vrinnevi Hospital
Other Study IDs: Dnr 2023-02252-01
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Inflammation; Genetic Predisposition to Disease
MeSH Terms: conditions — Atrial Fibrillation; Inflammation; Genetic Predisposition to Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective cohort: Prospective cohort measuring the previously described biomarkers.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling

SUMMARY:
Because of the high recurrence rates following electrical cardioversion and high morbidity in AF patients there is a need to explore prediction models for AF recurrence following ECV. Previous studies have primarily focused on high-sensitivity CRP (hsCRP), CRP, and IL-6, while other inflammatory indexes and gene scores might hold greater value.

This prospective cohort study is planning to include 182 patients with persistent atrial fibrillation, planned for electrical cardioversion, and >18 years at two medium-sized hospitals in Sweden. Blood samples will be collected prior to electrical cardioversion and at 7-, 30-, 90-, and 180-days follow-up. Atrial fibrillation recurrence will be evaluated at follow-up or upon patient request and diagnosed with 12-lead ECG.

An interim analysis will be conducted after more than 80 patients have been included. If the results from univariate and/or multivariable logistic regression on inflammatory markers and genetic expression regarding atrial fibrillation recurrence are significant, the study will be concluded.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation (ICD-10 I48.1)
* Age over 18 years

Exclusion Criteria:

* Autoimmune disease
* Inflammatory diseases
* Acute or chronic liver dysfunction
* Ongoing infectious diseases
* Thyroid disorders
* Any other conditions known to impact inflammatory activity (including medication use and hematological diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included patients aged 18 or older diagnosed with persistent atrial fibrillation (ICD-10 I48.1) scheduled for ECV. Inclusion took place from 2023-10-18 to 2025-06-01.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence of AF | During follow-up (post ECV, day 7, 30, 90, and 180)
  Recurrence of atrial fibrillation or atrial flutter recorded on 12-lead ECG or through pacemaker interpretation

SECONDARY OUTCOMES:
Fluctuations of biomarkers and gene expression during follow-up | During follow-up (post ECV, day 7, 30, 90, and 180)
  Change in biomarker level or expression of gene expressions during follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Medical department, Jönköping, Småland
  - Cardiology Clinic, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No